CLINICAL TRIAL: NCT03897244
Title: Efficacies of High-dose Dual Therapy With or Without Bismuth Versus Amoxicillin-metronidazole Bismuth Quadruple Therapy for First-line Helicobacter Pylori Eradication - A Prospective, Randomized, Comparative Study
Brief Title: Efficacies of HDDT With or Without Bismuth vs Amoxicillin-metronidazole BQT for First-line H Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201812129MINC
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; high dose dual therapy; bismuth high-dose dual therapy; bismuth quadruple therapy
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Proton Pump Inhibitors; Anti-Bacterial Agents; Bismuth; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-dose dual therapy (Experimental): group A - HDDT (rabeprazole 20 mg qid + amoxicillin 750 mg qid, for 14 days)
  Interventions: Drug: High-dose dual therapy (rabeprazole, amoxicillin)
- Bismuth High-dose dual therapy (Experimental): group B - Bis-HDDT (rabeprazole 20 mg qid + amoxicillin 750 mg qid + tripotassium dicitrate bismuthate 300 mg qid, for 14 days)
  Interventions: Drug: Bismuth High-dose dual therapy (rabeprazole, amoxicillin, tripotassium dicitrate bismuthate)
- Amoxicillin-Metronidazole Bismuth quadruple therapy (Active Comparator): group C - AM-BQT (rabeprazole 20 mg bid + tripotassium dicitrate bismuthate 600 mg bid + amoxicillin 1000 mg bid + metronidazole 500 mg tid, for 14 days)
  Interventions: Drug: Amoxicillin-Metronidazole Bismuth quadruple therapy

INTERVENTIONS:
Drug: High-dose dual therapy (rabeprazole, amoxicillin) — High-dose dual therapy (rabeprazole 20 mg qid + amoxicillin 750 mg qid, for 14 days)
  Other Names: Proton pump inhibitor, Rabeprazole, Pariet®; Antibiotics, Amoxicillin ,Amoxicillin®
  Arms: High-dose dual therapy
Drug: Bismuth High-dose dual therapy (rabeprazole, amoxicillin, tripotassium dicitrate bismuthate) — Bismuth-High-dose dual therapy (rabeprazole 20 mg qid + amoxicillin 750 mg qid + tripotassium dicitrate bismuthate 300 mg qid, for 14 days)
  Other Names: Proton pump inhibitor, Rabeprazole, Pariet®; Antibiotics, Amoxicillin ,Amoxicillin®; Colloidal Bismuth, Tripotassium dicitrate bismuthate, KCB®
  Arms: Bismuth High-dose dual therapy
Drug: Amoxicillin-Metronidazole Bismuth quadruple therapy — Amoxicillin-Metronidazole Bismuth quadruple therapy (rabeprazole 20 mg bid + tripotassium dicitrate bismuthate 600 mg bid + amoxicillin 1000 mg bid + metronidazole 500 mg tid, for 14 days)
  Other Names: Proton pump inhibitor, Rabeprazole, Pariet®; Antibiotics, Amoxicillin, Amoxicillin®; Antibiotics, Metronidazole, Flagyl®; Colloidal Bismuth, Tripotassium dicitrate bismuthate, KCB®
  Arms: Amoxicillin-Metronidazole Bismuth quadruple therapy

SUMMARY:
Up to know, three is few large-scale, randomized study prospectively and simultaneously comparing the efficacy, adverse effects and patient compliance of high-dose dual therapy (HDDT) with or without bismuth versus amoxicillin-metronidazole bismuth quadruple therapy (AM-BQT) as first-line regimens for H. pylori eradication.

The aims of this study are:

1. to compare the efficacy of HDDT with or without bismuth and AM-BQT as first-line regimens for H. pylori eradication;
2. to compare the patient adherence and adverse effects of these treatment regimens;
3. to investigate factors that may influence H. pylori eradication by these treatment regimens;
4. to identify the effect of H. pylori eradication on the evolution of ecosystem of microbiota, and inflammatory parameters.

DETAILED DESCRIPTION:
This prospective multicenter randomized comparative study will be conducted at the National Taiwan University Hospital(NTUH), NTUH Bei-Hu Branch, NTUH Hsin-Chu Branch, Buddhist Tzu Chi General Hospital, and Mennonite Christian Hospital in Hua-Lien City. Patients, aged >= 20, having H. pylori-positive chronic gastritis with/without peptic ulcers (duodenal or gastric ulcers) will be recruited. All undergo endoscopy with biopsy for rapid urease test, histology, and bacterial culture before treatment. If the patients did not receive anti-H. pylori therapy previously, these patients will be invited to enter this study for evaluating the efficacy of these 1st-line regimens.

A computed generated random numbers sequence will be blocked into three subgroups, say A, B, and C. After giving written informed consent, each patient will be randomly allocated, to one of three treatment groups:

group A - HDDT (rabeprazole 20 mg qid + amoxicillin 750 mg qid for 14 days);

group B - Bis-HDDT (rabeprazole 20 mg qid + amoxicillin 750 mg qid + tripotassium dicitrate bismuthate 300 mg qid, for 14 days);

group C - AM-BQT (rabeprazole 20 mg bid + tripotassium dicitrate bismuthate 600 mg bid + amoxicillin 1000 mg bid + metronidazole 500 mg tid , for 14 days);

All patients will be asked to complete a questionnaire and to record symptoms, drug consumption, and diet content daily during the treatment period. Post-treatment, the patients will be followed up at the Outpatients Clinic to investigate patient adherence and adverse effects of treatment. Four to eight weeks after termination of treatment, H. pylori infection status will be examined by the C13-urea breath test (UBT). The CYP2C19 genotype of each participant will be analyzed by the polymerase chain reaction-based restriction fragment length polymorphism (PCR-RFLP) method. A part of participants, at least 30 cases in each group, will be invited to join a follow-up program for one year for evaluating the changes or evolution of gut microbiota composition, metabolic product, parameters of inflammation and immune response.

ELIGIBILITY:
inclusion criteria: participants having H. pylori related chronic gastritis with/without peptic ulcers who are aged greater than 20 years old and are willing to received first-line eradication therapy.

Exclusion criteria:

1. pregnant or nursing woman;
2. serious concomitant illness and malignant tumor of any kind;
3. history of hypersensitivity to test drugs；
4. serious bleeding during the course of this ulcer;
5. previous gastric surgery;
6. receiving bismuth salts, proton pump inhibitors (PPIs), or antibiotics in the previous month.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
to compare the eradication rate of HDDT with or without bismuth and AM-BQT as first-line regimens for H. pylori eradication. | 5.5 years
  The eradication rates (efficacy) of these regimens will be evaluated by the results of C13-urea breath test.

SECONDARY OUTCOMES:
to compare the patient adherence and frequency of adverse effects of these treatment regimens. | 5.5 years
  The frequency of adverse events will be evaluated by the number of participant with adverse events and patient adherence will be evaluated by counting unused medication after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D.Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan